CLINICAL TRIAL: NCT02076022
Title: Adipose Stromal Cell Enriched Autologous Fat Grafting for Treating Pain at Amputation Sites: A Single Center Site, Prospective, Randomized, Pilot Outcomes Trial
Brief Title: AMP30: Autologous Fat Grafting, Amputation Sites Pain: Randomized
Acronym: AMP30
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J. Peter Rubin, MD (Other)
Responsible Party: Sponsor-Investigator, J. Peter Rubin, MD, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PRO12050147
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2019-08-22 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Wounded Warrior; Limb Shortening; Amputation
Keywords: Fat Grafting; Pain at amputation site; prosthetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard fat grafting (Active Comparator): Once harvested the aspirated fat tissue will be processed as standard graft material. It will be divided into small aliquots and centrifuged in a sterile rotor (3000 rpm for 3 minutes/1200g), and top fluid oil layer from the fat tissue fractions were removed, and transferred into 1ml syringes and injected into the amputation stump. This graft preparation will be performed in the operating room. Standard fat graft material will serve as a control treatment and will be injected into limb using specialized injection cannulas
  Interventions: Procedure: Standard fat graft
- Enhanced Fat Grafting (Experimental): Approximately 60 cc of lipoaspirate will be collected from the subject to be processed with the Tissue Genesis Cell Isolation System™ (CIS) to yield approximately 35cc of Stromal Vascular Fraction (SVF).Once harvested the aspirated fat will then be divided into two portions: one portion will be processed as standard graft material (standard/control graft) while the other portion will be used in a processing step that concentrates the adipose stromal cells.
  The aspirated fat processed as standard graft material will be divided into small aliquots and centrifuged in a sterile rotor (3000 rpm for 3 minutes/1200g), and allowed to decant before separating the fluid and oil layers from the fat tissue fractions, and transferred into 50 ml syringes. This graft preparation will be performed in the operating room.
  Interventions: Device: Enhanced Fat Grafting

INTERVENTIONS:
Device: Enhanced Fat Grafting — The stromal vascular fraction (SVF) cell suspension (device output) will be processed using the Tissue Genesis Cell Isolation System™
  The Standard graft material and the stromal vascular fraction cells will be mixed and subsequently injected into the amputated stump at a concentration of 2.0 - 3.0 x 10 6 stromal vascular cells/ml of injected fat graft to each site. The volume of each injected fat graft will depend on the volume requirements for each injured extremity.
  To manually combine the standard fat graft material and the SVF suspension (device output), each of the syringes will be connected via luer to luer lock. The contents of the lipoaspirate syringe are transferred to the SVF syringe and the cell suspension will be injected slowly back and forth between the two (2) syringes. The final 1 mL SVF-fat graft syringe is now considered cell-enriched and ready for injection into the subject.
  Other Names: Tissue Genesis Cell Isolation System™ (CIS)
  Arms: Enhanced Fat Grafting
Procedure: Standard fat graft — Aspirated fat tissue will be processed as standard graft material. It will be divided into small aliquots and centrifuged in a sterile rotor (3000 rpm for 3 minutes/1200g), and top fluid oil layer from the fat tissue fractions were removed, and transferred into 1ml syringes and injected into the amputation stump. This graft preparation will be performed in the operating room. Standard fat graft material will serve as a control treatment and will be injected into limb using specialized injection cannulas
  Arms: Standard fat grafting

SUMMARY:
We propose a prospective, randomized clinical study to assess the efficacy of minimally invasive autologous fat transfer addressing pain and poor prosthetic fit at amputation sites.

DETAILED DESCRIPTION:
We hypothesize that autologous fat grafting can provide a minimally invasive therapy facilitated by enabling technology of specialized instrumentation to effectively mitigate pain syndromes at amputation sites, by introducing volume stable subcutaneous tissue over bony prominences and peripheral nerve trunks, thereby avoiding surgical revisions and preserving limb length.

We further hypothesize that enriching the fat graft with autologous adipose stromal cells utilizing the Tissue Gensis Cell Isolation System (CIS), a regenerative medicine approach, will lead to improved retention of the fat graft over time and result in a more favorable outcome.

Specific Aims:

1. Treat painful amputation sites in 30 patients with fat grafting to provide additional subcutaneous tissue padding over bony structures and nerve trunks. Limb anatomy and healing of the graft over time, along with stability/persistence of the new tissue, will be assessed by high resolution CT scanning with 3D reconstruction. Patients will be followed for 24 months after treatment to define long term outcomes. The primary outcome measures will be pain at the amputation site and improved ability to tolerate a prosthesis. Patients will be randomized to receive either standard fat grafting (15 patients)or cell enriched fat grafting (15 patients). Patients will be enrolled who have pain at an amputation site that limits function and/or interferes with the ability to use a prosthesis.
2. Assess biologic properties of the cells within the fat graft and correlate with clinical outcomes. This will include adipose stem cell yield per volume of fat tissue, cell proliferation, capacity for adipogenic differentiation, lipolysis, and cell sub-population analysis by multiparameter flow cytometry. Results of these assays will be correlated with graft volume retention to search for predictors of good clinical outcome that are related to variation on adipose biology between subjects.
3. Measure quality of life in patients before and after autologous fat grafting using validated psychosocial measures. This will include, among other tools, SF 36, the Beck inventory, and instruments designed for assessing limb function.

Study Design:

Single center site, prospective, randomized, pilot outcomes study with treatment performed at the University of Pittsburgh.

The primary outcome measurements will be: 1) fat graft retention at the amputation site; and 2) improved ability to tolerate a prosthetic device. This study will examine if fat grafting with cell enrichment using the Tissue Gensis Cell Isolation System, (CIS) will demonstrate increased fat retention and decreased pain compared to standard fat grafting alone.

Clinical Impact:

This study will significantly impact military trauma care by validating a minimally invasive cell based technique for alleviating pain at amputation sites and improving function with a prosthesis. Importantly, the goal will be reached without invasive surgery, increased risk, and a prolonged recovery. Given the high amputation rate in the current conflicts, this work is highly relevant to the care of the wounded warrior. A major goal of this study will be to transfer the techniques and knowledge gained to physicians throughout the Department of Defense healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older and able to provide informed consent
* Has an amputation with pain that limits the fitting and use of a prosthesis, despite maximal attempts to refit the prosthesis and/or change the design of the prosthesis and/or Have an amputation with pain that limits the use of an assistive device(s) despite maximal attempts to change the design of use of the device
* Be at least 3 months post-injury or post-surgery (from trauma procedures) so that acute edema is resolved
* Soft tissue deficiencies are noted at amputation stump and are covered by intact skin
* Willing and able to comply with follow up examinations, including radiographic studies
* Subjects who are, in the opinion of the Investigator, able to understand the study, comply with the study design and are willing to return to the clinic for all the research required follow-up visits
* Subjects with residual limb problems including upper and lower limb loss, and/or individuals with partial hand, partial foot and more proximal injuries.
* Subjects with Intolerability that may include appropriate soft tissue padding, soft tissue coverage, or pain that doesn't allow the consistent wearing of a prosthetic socket. (This may include excessive pain, inability to achieve adequate suspension of prosthesis on the individual, continual skin breakdown, excessive pressure/shear on skin, soft tissue, nerves, scars, etc.) and/or Subjects with Intolerability that limits use of an assistive device(s) that aid mobility of daily living activities involving the functional use of affected limb.
* Subjects who are unable to consistently wear a prosthetic socket must have received a minimum of 3 months of unsuccessful prosthetic fitting trials. This will include a minimum of at least 5 different socket adjustments. This can include re-casting the residual limb, providing pressure relieves within the socket, changing the alignment of the prosthetic components to alter ground reactive forces, and adding padding to pressure sensitive areas. Likewise, subjects using assistive devices must have received a minimum of 3 months of unsuccessful assistive device adjustments. This information pertaining to the history of prosthetic fit attempts may be received from referral physician, prosthetics and/or orthotics direct report and/or subject self-report and/or medical record review.
* Subjects should have an approximate range of the defect volume between 5cc to as much as 300cc. if the defect is a very local soft tissue deficiency over a pressure point. (The volume of the defect correlates with moderate or severe intolerability of the prosthesis)
* Subjects must have a current relationship with a prosthetist and/or Assistive device Technician.
* Subjects who have a history of cancer to an affected limb that results in a surgical amputation maybe eligible.
* Subjects who have a history of embolus to the affected limb that results in surgical amputation maybe eligible

Exclusion Criteria:

* Age less than 18 years
* Patient has inability to provide informed consent process.
* Amputated limb area intended for treatment has open wounds or tunneling
* Active drainage or active infection unresolved with one course of antibiotic treatment
* Active infection anywhere in the body
* Diagnosed with cancer within the last 12 months and /or presently receiving chemotherapy or radiation treatment
* Known coagulopathy symptoms /diagnosis
* Systemic disease that would render the fat harvest and injection procedure, along with associated anesthesia, unsafe to the patient (e.g., scleroderma, lupus, vasculatures, collagen disease etc.)
* Pregnancy
* History of Diabetes Mellitus
* History of severe peripheral arterial disease
* Subjects with an Axis I DSM-IV diagnosis (e.g., Schizophrenia, Bipolar disorder) who are found to be clinically (i.e. medically) unstable at baseline. Individuals who manifest either: 1) evidence of currently active alcohol or psychoactive drug abuse or dependence on the SCID interview, or 2) a GAF score of 40 or lower due to any acute psychiatric symptomatology (e.g. suicidality, psychosis, severe depression or mania) will be reviewed by the Co-I for Psychosocial Assessment with the PI for determination of possible medical instability. Final determination of medically unstable status will be made by the PI on the basis of overall medical status and appropriateness for medical procedures; the patient may be considered ineligible for study participation per the Physician's discretion.
* Subjects with abnormal blood biochemistry or any other abnormal laboratory finding considered clinically significant in that it would deem the subject inappropriate for surgical procedures. This criterion will help to exclude subjects with severe nutritional deficiency, anemia, coagulopathy, renal and liver dysfunction, diabetes, and peripheral vascular disease, as determined by the investigator (i.e. CBC with Differential, platelets, comprehensive metabolic panel to include electrolytes, bun/creatinine, liver function test and coagulation tests). As general safety measures, we will exclude patients with lab values listed below: Hct less than 30% INR greater than 1.8 Creatinine greater than 2.0 Liver function tests (ALT, AST, Bilirubin) greater than 2 times upper limit Albumin- Less than 2.0 Platelets less than 70
* Subjects who per the clinical discretion of the investigator, would not be appropriate for the study. (e.g. a potential medication and/ or medical diagnosis that is not captured in above exclusion, but which could render the subject's participation in the study unsafe, or would have an adverse effect on fat metabolism or fat healing).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-04-08 (Actual); Primary Completion 2018-07-18 (Actual); Study Completion 2019-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Rubin, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
It is the Principal Investigator's intention to make subject de-identified information available to secondary investigators after all research study testing has been completed. These associated subject information will not include subject identifiers.

REFERENCES:
- See also: University of Pittsburgh Department of Plastic Surgery — http://www.plasticsurgery.pitt.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard Fat Grafting | Enhanced Fat Grafting
Started | 7 | 3
Completed | 5 | 3
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Fat Grafting | Enhanced Fat Grafting | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (13.0) | 46.4 (18.1) | 49.9 (16.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 7 | 2 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Autologous Fat Transfer at Pain Modulation at Respective Amputation Sites
Description: Assess the efficacy of minimally invasive autologous fat transfer at the amputation sites and the modulation of pain at the respective sites
  Compare two minimally invasive techniques as an alternative to invasive operations, with the understanding that this therapy does not preclude more invasive procedures in the future. We further hypothesize that enriching the fat graft with autologous adipose stromal cells utilizing the Tissue Genesis Cell Isolation System (CIS), a regenerative medicine approach, will lead to improved retention of the fat graft over time and result in a more favorable outcome.
  Subjects reported pain on a scale of 0-5 where 5 was the worst pain and 0 was no pain.
Time Frame: 2 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Standard Fat Grafting | Enhanced Fat Grafting
Number analyzed (Participants) | 7 | 3
score on a scale | 1.3 (1) | 0 (0)

2. Secondary Outcome: Cell Yield
Description: To assess biologic properties of the cells within the fat graft, we evaluated adipose stem cell viability by multiparameter flow cytometry.
Time Frame: day 0
Population: participant discrepancy due to subject withdrawal from study
Measure: Mean (Standard Deviation); unit: percentage of SVF cell viability
Arm/Group | Standard Fat Grafting | Enhanced Fat Grafting
Number analyzed (Participants) | 6 | 2
percentage of SVF cell viability | 69.9 (31.8) | 82.7 (3.6)

3. Secondary Outcome: Number of Participants With Clinically Significant Levels of Depression on the Patient Health Questionnaire-9 (PHQ-9)
Description: Measure quality of life in patients before and after autologous fat grafting using validated psychosocial measures. This will evaluate using instruments designed for assessing depression including the Patient Health Questionnaire-9 (PHQ-9) which is a tool to screen, diagnose, monitor, and measure the severity of depression.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Fat Grafting | Enhanced Fat Grafting
Number analyzed (Participants) | 5 | 3
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Standard Fat Grafting | Enhanced Fat Grafting
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 7/7 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard Fat Grafting (N=7) | Enhanced Fat Grafting (N=3)
Bruising at donor site (Surgical and medical procedures) | 7 (7) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/22/NCT02076022/Prot_SAP_000.pdf
  • Informed Consent Form (2014-01-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT02076022/ICF_001.pdf